CLINICAL TRIAL: NCT03649373
Title: The Noergaard Technique, a Simple and Non-traumatic Method for Reduction of Anterior Shoulder Dislocations
Brief Title: The Noergaard Technique for Anterior Shoulder Dislocation
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Nikolaj Erin-Madsen, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: Noergaard Study
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Anterior Shoulder Dislocation
Keywords: Shoulder; Dislocation; Noergaard; Reduction
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ED Patients: We retrospectively reviewed patient charts of all patients admitted for shoulder dislocation at the ED at Copenhagen University Hospital Hvidovre between January 1st 2014 and December 31st 2014. A total of 151 patients' charts were reviewed.
  Interventions: Procedure: Noergaard technique

INTERVENTIONS:
Procedure: Noergaard technique — The patient is placed standing in an upright position in front of the rail on a hospital bed. Legs should be stretched with a wide well balanced stance. The patient is then instructed to bend forwards, resting the forehead on the back of the non-affected forearm, which is put on the rail. The affected arm should now be relaxed and stretched, hanging straight down toward the floor. The patient is then instructed to attempt to relax and make pendular and circular motions with the affected arm hanging down. Successful reduction occurs when sufficient muscle relaxation allows the humeral head to reposition to its natural position in the glenoid fossa. Often the patient will experience a popping sensation when the shoulder is reduced.

SUMMARY:
In this paper we describe and evaluate the results of the Noergaard technique through a retrospective analysis of patients admitted and treated for anterior shoulder dislocation at the ED of Copenhagen University Hospital Hvidovre, Denmark, in a 1-year period.

DETAILED DESCRIPTION:
Introduction

In this article the investigators describe the Noergaard technique for reduction of anterior shoulder dislocations. This is an atraumatic reduction method that has proven successful through several years of practice. The investigators describe and evaluate the results of this technique through a retrospective analysis of patients admitted and treated for anterior shoulder dislocation at the emergency department (ED) of Copenhagen University Hospital Hvidovre, Denmark, in a 1-year period.

Methods

In the Noergaard technique the patient is placed standing bend over forwards in front of the rail on a hospital bed, resting the forehead on the back of the non-affected forearm, which is put on the rail. The affected arm should now be relaxed and stretched, hanging straight down toward the floor. The patient is then instructed to attempt to relax and make pendular and circular motions with the affected arm hanging down.

ELIGIBILITY:
Inclusion Criteria:

- Patients have had a closed shoulder reduction performed at the emergency center of Hospital of Hvidovre between 1st of January 2014 and the 31st of December 2014.

Exclusion Criteria:

* Patients with diagnosed severe arthrosis in the shoulder joint.
* Patients with malignancy in the humerus or scapula.
* Patients who have had a Total Shoulder Arthroplasty performed at the same side as the lunation.
* Patients with more than four previous shoulder reductions performed.
* Patients who have undergone operations on the same shoulder, but at different hospitals.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is chosen from the criteria that patients have had a closed shoulder reduction performed at the emergency center of Hospital of Hvidovre between 1st of January 2014 and the 31st of December 2014.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Successful shoulder reduction after anterior shoulder dislocation. | 30 min.
  Successful shoulder reduction occurs when sufficient muscle relaxation allows the humeral head to reposition to its natural position in the glenoid fossa.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj Erin-Madsen, MD, Study Director — Copenhagen University Hospital of Hvidovre

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan.

REFERENCES:
- [Background] Canale ST, Beaty JH, Phillips BB. Recurrent dislocation in Canley and Beaty: Campbell's Operative Orthopaedics. 11th edition. Vol. 45. Philadelphia: Mosby Elsevier; 2007. pp. 2677-83.
- [Background] Beattie TF, Steedman DJ, McGowan A, Robertson CE. A comparison of the Milch and Kocher techniques for acute anterior dislocation of the shoulder. Injury. 1986 Sep;17(5):349-52. doi: 10.1016/0020-1383(86)90161-0. PMID 3533776
- [Background] Manes HR. A new method of shoulder reduction in the elderly. Clin Orthop Relat Res. 1980 Mar-Apr;(147):200-2. PMID 7371296
- [Background] Plummer D, Clinton J. The external rotation method for reduction of acute anterior shoulder dislocation. Emerg Med Clin North Am. 1989 Feb;7(1):165-75. PMID 2917505
- [Background] Marinelli M, de Palma L. The external rotation method for reduction of acute anterior shoulder dislocations. J Orthop Traumatol. 2009 Mar;10(1):17-20. doi: 10.1007/s10195-008-0040-4. Epub 2009 Jan 8. PMID 19384630
- [Background] MILCH H. The treatment of recent dislocations and fracture-dislocations of the shoulder. J Bone Joint Surg Am. 1949 Jan;31A(1):173-80. No abstract available. PMID 18106759
- [Background] Canales Cortes V, Garcia-Dihinx Checa L, Rodriguez Vela J. Reduction of acute anterior dislocations of the shoulder without anaesthesia in the position of maximum muscular relaxation. Int Orthop. 1989;13(4):259-62. doi: 10.1007/BF00268508. PMID 2599702
- [Derived] Erin-Madsen N, Ban I, Thomsen MG, Noergaard J, Tengberg PT. The Noergaard technique is a non-traumatic method for reduction of anterior shoulder dislocation. Dan Med J. 2021 Mar 17;68(4):A06200422. PMID 33829988